CLINICAL TRIAL: NCT01683591
Title: Dysphagia Screening in Acute Stroke Using High-resolution Impedance Manometry (DASH); Its Implication to Diet Decision and Clinical Outcome
Brief Title: Dysphagia Assessment in Acute Ischemic Stroke Using High-resolution Manometry
Acronym: DASH
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Joongseok Kim, Associate Professor, The Catholic University of Korea
Other Study IDs: 060613
Record Dates: First submitted 2012-09-04; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Ischemic Stroke
Keywords: Acute stroke; Dysphagia; High-resolution manometry
MeSH Terms: conditions — Ischemic Stroke; Stroke; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High-risk aspiration group: Among the consecutive stroke patients, categorized to high-risk group in the patient (1) was not on alert mentality (from drowsy to comatose mentality), (2) was not able to sit upright or control his/her head, and (3) failed to pass indirect water swallow test.
- Low-risk aspiration group: Patents without oropharyngeal neurologic signs
- Intermediate-risk aspiration group: If any one of following was positive, categorized to intermediate-risk group; (1) dysarthria, (2) motor aphasia, (3) inability to close and open lips or (4) facial weakness, (5) tongue deviation or (6) uvula deviation, (7) loss of gag reflex, and (8) inability to cough voluntarily.
  Interventions: Procedure: High-resolution impedance manometry test

INTERVENTIONS:
Procedure: High-resolution impedance manometry test — The test was performed as general guideline for high-resolution impedance manometry test. The parameter was obtained and analyzed using the Chicago classification for the liquid swallows with Takasaki's modification for pharyngeal function monitoring. Swallowing pattern and aspiration risk were defined using real-time assessment of high-resolution impedance manometry test.
  Other Names: ManoScan360 and ManoScanZ (Sierra Scientific Instruments, Los Angeles, CA).
  Groups: Intermediate-risk aspiration group

SUMMARY:
Dysphagia occurs relatively commonly in patients with acute stroke, and can lead to aspiration pneumonia and malnutrition. By using the stroke registry of our hospital, we will evaluate the feasibility and usefulness of Dysphagia screening in Acute Stroke using High-resolution impedance manometry (DASH). The hypothesis tested in this study is that high-resolution impedance manometry (HRiM) can provide the clinical efficacy to evaluate dysphagia and the diet plan in acute stroke patients.

DETAILED DESCRIPTION:
The hypothesis tested in this study was that high-resolution manometry can provide the clinical efficacy to evaluate dysphagia and the diet plan in acute stroke patients. By using of stroke registry of our hospital, we assessed feasibility and usefulness of Dysphagia screening in Acute Stroke using High-resolution impedance manometry in patients with acute stroke.

The registry had the contents of two evaluation steps; the first step was the process to identify the patients with risk of possible aspiration and the second step was for detection of silent aspirators.

Firstly, the patient was interviewed regarding difficulties with food intake, chewing and swallowing, and the neurological signs were confirmed by two independent neurologists. After then, the patients were stratified into three aspiration risk group and controlled by proper diet program. Finally the emergence of aspiration pneumonia was observed.

ELIGIBILITY:
Inclusion Criteria: New stroke lesion should be present in MRI which compatible with clinical history and neurologic examination and patients with onset <= 48 hours.

Exclusion Criteria:

1. hyperacute stroke receiving thrombolytic therapy
2. symptom onset > 48 hours
3. patients who died in the incipient stage of acute stroke
4. neurological deterioration (increase in NIHSS ≥ 4)
5. transient ischemic attack
6. history of prior stroke and dysphagia
7. other neurological diseases causing oropharyngeal dysphagia, such as Parkinsonism, dementia, and neuromuscular disorders
8. history of cranial neurosurgery
9. prior or current structural lesions causing oropharyngeal dysphagia,
10. pulmonary diseases such as chronic obstructive pulmonary disease or current pneumonia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute ischemic stroke patients at neurology department from April 2009 to November 2009 were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2009-04; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Improvement of diet program | Cases were followed for the duration of hospital stay, an average of 2 weeks.
  All patients with dysphagia received swallowing rehabilitation training and were guided as per National Dysphagia Diet level or nasogastric tube feeding. These patients were monitored in terms of the improvement of dietary program (e.g., From nasogastric tube feeding to step 4 dysphagia diet).
Occurrence of aspiration pneumonia | Cases were followed for the duration of hospital stay, an average of 2 weeks.
  All patients were monitored in terms of development of aspiration pneumonia. Aspiration pneumonia was defined as typical clinical signs (fever, sputum etc.) and chest radiographic findings (X-ray and computed tomography etc.).

SECONDARY OUTCOMES:
Overall satisfaction measurement regarding program | 1 month after study enrollment
  The patients also answered as visual analogue scales that measured their level of overall satisfaction regarding improvement of their symptoms with the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Joongseok Kim, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea